CLINICAL TRIAL: NCT05418244
Title: Inhaled Isopropyl Alcohol for the Treatment of Nausea in a Pediatric Emergency Department: A Open Label, Randomized Controlled Clinical Trial
Brief Title: Inhaled Isopropyl Alcohol for Treatment of Nausea
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Susana Ruano, Pediatric Emergency Medicine Fellow, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00005944
Record Dates: First submitted 2022-06-01; First posted 2022-06-14 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Vomiting; Nausea; Children, Only
MeSH Terms: conditions — Vomiting; Nausea | interventions — Ethanol; Ondansetron

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inhaled Isopropyl Alcohol (Experimental): If the subject is assigned to receive the isopropyl alcohol pad group, an isopropyl alcohol pad (Covidien Webcol 2 ply prep pad, saturated with 70% isopropyl alcohol) will be given to the subject, or the legal guardian. The alcohol pad will be held 1-2 cm under the subject's nares, the subject will be instructed to take deep breaths, inhaling through the nose as frequently as needed during the Emergency Department (ED) stay.
  Interventions: Other: Inhaled Isopropyl Alcohol
- Oral Ondansetron (Active Comparator): If the subject is assigned to receive ondansetron treatment, subject will be provided with 4 mg ondansetron oral disintegrating tablet (ODT) for treatment.
  Interventions: Drug: Oral Ondansetron
- Inhaled Placebo (Placebo Comparator): If the subject is assigned to receive the inhaled placebo, a normal saline pad (Hygea sterile saline wipe) will be given to the subject or the legal guardian. The saline wipe will be held under the subject's nares, the subject will be instructed to take deep breaths, inhaling through the nose as frequently as needed.
  Interventions: Other: Inhaled Placebo

INTERVENTIONS:
Other: Inhaled Isopropyl Alcohol — Isopropyl alcohol pad (Covidien Webcol 2 ply prep pads, saturated with 70% isopropyl alcohol) held 1-2 cm under the subject's nares
  Other Names: Webcol
  Arms: Inhaled Isopropyl Alcohol
Drug: Oral Ondansetron — 4 mg oral disintegrating ondansetron tablet once
  Other Names: Zofran
  Arms: Oral Ondansetron
Other: Inhaled Placebo — Normal saline pad (Hygea sterile saline wipe) held 1-2 cm under the subject's nares
  Other Names: Inhaled Normal Saline'
  Arms: Inhaled Placebo

SUMMARY:
To determine the efficacy of inhaled isopropyl alcohol in treating nausea/vomiting among pediatric patients compared with the conventional ondansetron, or placebo treatment in a tertiary care pediatric emergency department.

DETAILED DESCRIPTION:
I. Obtaining consent Our study personnel will approach the treating physician in the ED once a patient is suspected to be eligible for the study. The physician will determine patient's eligibility by using the screening sheet. If a patient meets all study inclusion and exclusion criteria, our study personnel will approach the legal guardian/patient in the private patient room and introduce the study to them. Enough time will be given to the patient and their legal guardian to allow them review and understand the consent/assent. All questions will be answered before obtaining the consent. Once the consent/assent is obtained from the legal guardian and participant, our study personnel will keep the treating physician and bedside nurse posted about the enrollment.

II. Randomization of subject

There will be three arms of this study:

1. Conventional oral ondansetron (Zofran) treatment group,
2. Inhaled isopropyl alcohol treatment group,
3. Inhaled normal saline (placebo) group. After obtaining informed consent, the patients will be randomized into one of the three groups following a randomization table created by a statistician.

Whichever intervention is randomly selected will be used to treat the subject. Our research team member will notify the treating physician and the bedside RN about the assignment.

If the subject is assigned to receive ondansetron treatment, subject will be provided with 4 mg ondansetron oral disintegrating tablet (ODT) for treatment.

If the subject is assigned to receive the isopropyl alcohol pad group, an isopropyl alcohol pad (Covidien Webcol 2 ply prep pads, saturated with 70% isopropyl alcohol) will be given to the subject, or the legal guardian . The alcohol pad will be held 1-2 cm under the subject's nares, the subject will be instructed to take deep breaths, inhaling through the nose as frequently as needed during the ED stay.

If the subject is assigned to receive the inhaled placebo, a normal saline pad (Hygea sterile saline wipe) will be given to the subject or the legal guardian. The saline wipe will be held under the subject's nares, the subject will be instructed to take deep breaths, inhaling through the nose as frequently as needed.

For those subject who receives normal saline or alcohol pad treatment, if their vomit/nausea symptoms has not improvement after 30 minutes post intervention, they may receive Zofran treatment in the ED.

III. Data collection A paper data collection form will be used to collect data in the ED, which is attached with this submission. Patient ID sticker with name, MRN, FIN, and DOB will be placed on the data form. This data form will be completed by the ED research assistant. The completed data form as well as the signed informed consent document will be placed in a locked study data box in the ED. The study coordinator will collect these documents from the ED periodically, and transfer the documents to the UBMD Pediatrics Department Research Office (5th Floor Conventus, 1001 Main St, Buffalo, NY 14203). All paper documents will be stored in locked file cabinet in the office.

Two databases will be created for this study, the Subject Database and the PHI database. Subject identifiable information will be entered in the PHI database, which include: MRN, FIN, and DOB. All other data elements will be entered in the Subject Database. Certain PHI e.g. ED visit/discharge date, study intervention administration date will also be entered in the Subject database for the convenience of data analysis. A unique study ID will be assigned to each subject, this ID number will be used as the code key to link the paper data form, Subject Database and PHI database. Both databases will be saved in study coordinator's password protected UPA online drive, the PHI database will be double secured by a code.

Data Collection:

1. Demographic data: Patient age, sex, race, and ethnicity
2. Baxter Animated Retching Faces nausea score at: Baseline (prior to intervention), 10 minutes post-intervention, 30 minutes post-intervention, and at ED discharge.

   The 10 minute post-intervention timepoint was selected because prior research in adult post-operative patients has shown that inhaled isopropyl alcohol significantly improved nausea on surveys conducted 5, 10, and 15 minute after inhalation.6 The 30 minute post-intervention timepoint was selected because the onset of action for ondansetron oral disintegrated tablet is within 30 minutes.132 We will reassess nausea symptoms at ED discharge to account for any anti-emetic benefit that may have only be transient.
3. ED clinical information about vomiting and apparent aspiration
4. Patient/caregiver perceived side effects of treatment
5. Satisfaction scores: From both the bedside nurse and the patient's caregiver
6. Cross-over information: Did the patient use a treatment other than the assigned treatment (e.g. if the patient was in the inhaled isopropyl alcohol group, did they cross-over into the ondansetron ODT group)
7. ED discharge information: Length of stay, patient disposition and discharge diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patients with a chief complaint of nausea or vomiting
* Ages 7-178 years, both sexes
* Weight ≥ 15 kg
* Baxter Animated Retching Faces (BARF) nausea severity score ≥ 4/10

Exclusion Criteria:

* 1. Require IV access
* Inability to breathe in/out through the nose
* Anosmia (self- or parental report)
* Allergy to isopropyl alcohol or ondansetron
* Current or history of alcohol abuse
* Inability to communicate feeling nauseous
* Inability to follow directions regarding taking deep breaths through the nose
* Known prolonged QT interval
* Pregnancy
* Received antiemetics within the last 8 hours
* Currently taking apomorphine

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Nausea Score at 30 Minutes | 30 minutes post-intervention as compared to baseline
  Baxter Animated Retching Faces nausea score, 0-10 with higher score meaning worse nausea
Change in Nausea Score at 10 Minutes | 10 minutes post-interventnon as compared to baseline
  Baxter Animated Retching Faces nausea score, 0-10 with higher score meaning worse nausea
Change in Nausea Score at Discharge | At ED discharge (assessed up to 10 hours) as compared to baseline
  Baxter Animated Retching Faces nausea score, 0-10 with higher score meaning worse nausea

SECONDARY OUTCOMES:
Vomiting | From intervention to time of ED discharge (assessed up to 10 hours)
  Number of episodes of vomiting post-intervention
Parent/Caregiver Satisfaction | At time of ED discharge (assessed up to 10 hours)
  Patient's parent/caregiver satisfaction score (very dissatisfied, dissatisfied, neutral, satisfied, very satisfied)
Nurse Satisfaction in Ease of Administering the Treatment | At time of ED discharge (assessed up to 10 hours)
  Patient's bedside nurse satisfaction score (very difficult, somewhat difficult, neutral, somewhat easy, very easy)
Length of Stay | From arrival to time of ED discharge (assessed up to 10 hours)
  Length of patient's stay in the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Alana Koehler, MD, Principal Investigator — SUNY Buffalo; Heather Territo, MD, Study Director — SUNY Buffalo
Locations (1):
- Oishei Children's Hospital, Buffalo, New York, United States